CLINICAL TRIAL: NCT00073840
Title: An Efficacy and Safety Study of Levalbuterol, Racemic Albuterol and Placebo in Subjects Twelve Years of Age and Older With Asthma
Brief Title: Study of Levalbuterol, Racemic Albuterol and Placebo in Subjects Twelve Years of Age and Older With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 051-355
Record Dates: First submitted 2003-12-09; First posted 2003-12-11 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: levalbuterol; asthma; bronchoconstriction; adolescent; adult
MeSH Terms: conditions — Asthma | interventions — Levalbuterol; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Active Comparator): Levalbuterol 90 ųg QID (manufacturing site A or B)
  Interventions: Drug: levalbuterol
- II (Active Comparator): Racemic Albuterol 180 ųg QID
  Interventions: Drug: levalbuterol
- III (Placebo Comparator): Placebo QID
  Interventions: Drug: levalbuterol

INTERVENTIONS:
Drug: levalbuterol — * Levalbuterol 90 ųg QID (manufacturing sites A or B);
  * Racemic Albuterol 180 ųg QID;
  * Placebo QID
  Other Names: Xopenex HFA (levalbuterol tartrate)Inhalation Aerosol

SUMMARY:
The primary objective of this study is to investigate the efficacy of levalbuterol 90 ug (2 actuations, 45 ug each) versus placebo (2 actuations) in the treatment and prevention of bronchoconstriction in adolescent and adult subjects with asthma, with all treatments administered 4 times a day (QID).

DETAILED DESCRIPTION:
A double-blind, randomized, placebo- and active-controlled, multicenter, parallel-group trial of levalbuterol in subjects 12 years of age and older with asthma. Study participation will include one 1-week single-blind placebo run-in and an 8-week, randomized,double-blind, active-treatment period with four treatment groups. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Must give written informed consent (IC) prior to participation in the study. For subjects 12 - 17 years of age, the IC must be signed parent or legal guardian. Females must sign the Women of Childbearing Potential Addendum
* Be willing and able to comply with the study procedures and visit schedules
* Male or female, at least 12 years of age
* Females 12-60 years of age must have a negative serum pregnancy test at Visit 1 (V1)
* Women of child bearing potential must be using an acceptable method of birth control
* Must have a documented diagnosis of asthma for a min. of 6 mos. prior to V1
* At V1, the subject must demonstrate a baseline FEV1 within >45% and <75% of predicted for their height, age, gender, and race
* Following abstention from medications used to treat asthma, subject must demonstrate >12% reversibility of airflow obstruction within 15-30 min. following inhalation of 180 µg (2 actuations, 90 µg ea.) of racemic albuterol MDI
* Must have stable baseline asthma and have been using a B-adrenergic agonist, and/or anti-asthma anti-inflammatory medication, and/or OTC asthma medication for at least 6 mos. prior to V1
* Must be in good health with the exception of their reversible airways disease and not suffering from any chronic condition that might affect their respiratory function
* Must have a chest X-ray that is not diagnostic of pneumonia, atelectasis, pulmonary fibrotic disease, pneumothorax, chronic obstructive pulmonary disease, etc.
* Must be able to complete the diary cards and medical event calendars reliably on a daily basis and demonstrate how to use the MiniWright PEF meter

Exclusion Criteria

* Subject who is expected to require any disallowed medications
* Female subject who is pregnant or lactating
* Subject who has participated in an investigational drug study within 30 days prior to V1, or who is currently participating in another clinical trial
* Schedule prevents him or her from taking the first daily dose of study medication and/or starting study visits before 9AM
* Subject who has travel commitments during the study that would interfere with trial measurements or compliance or both
* Subject who has a history of hospitalization for asthma within 45 days prior to V1, or who is scheduled for in-patient hospitalization during the trial
* Have a known sensitivity to levalbuterol or racemic albuterol, or any of the excipients contained in any of these formulations
* Subject using any prescription drug with which albuterol sulfate administration is contraindicated
* Subject with currently diagnosed life-threatening asthma
* Subject with clinically significant abnormalities that may interfere with the metabolism or excretion of the study drug
* Have a history of cancer (exception: basal cell carcinoma in remission)
* Have hyperthyroidism, diabetes, hypertension, cardiac diseases, or seizure disorders not well controlled by medication or that may interfere with the successful completion of this protocol
* Have a history of substance or drug abuse within 12 mos. preceding V1 or a positive urine drug screening at V1
* Have greater than 10 pack year history of cigarette smoking or use of any tobacco products within 6 mos. of V1
* Have a documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis
* Have suffered from a clinically significant upper or lower respiratory tract infection in the 2 weeks prior to V1
* Have any clinically significant abnormal laboratory values
* Have a clinically significant abnormal 12-lead ECG that may jeopardize the subject's ability to complete study
* Subject who is a staff member or relative of a staff member

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2002-12; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
FEV1 (peak percent change from pre-dose averaged over the double-blind period). | 8 weeks

SECONDARY OUTCOMES:
--FEV1 [area under the % change from pre-dose FEV1 curve] and FEV1 [area under the % change from study baseline FEV1 curve] | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Hanrahan, M.D., Study Chair — Sumitomo Pharma America, Inc.
Locations (54):
- United States (54):
  - Allergy & Asthma Center, LLC, Oxford, Alabama
  - Alta Clinical Research, Tucson, Arizona
  - Integrated Research Group, Corona, California
  - Radiant Research, Inc., Encinitas, California
  - Allergy & Asthma Specialists Medical Group, Huntington Beach, California
  - Asthma, Allergy & Respiratory Care Center, Long Beach, California
  - Allergy Research Foundation, Inc., Los Angeles, California
  - Madera Family Medical Group, Madera, California
  - Southern California Research, Mission Viejo, California
  - Comprehensive Allergy Services, Oakland, California
  - Clinical Trials of Orange County, Orange, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy & Asthma Medical Group & Research Center, San Diego, California
  - Allergy & Asthma Assoc. of Santa Clara Valley Research Center, San Jose, California
  - West Coast Clinical Trials, Signal Hill, California
  - Allergy & Asthma Medical Group of Diablo Valley, Inc., Walnut Creek, California
  - 1st Allergy & Asthma Clinical Research Ctr, Thornton, Colorado
  - Watts Medical Research, Barnesville, Georgia
  - The Allergy & Asthma Clinical Research Center, Conyers, Georgia
  - Aeroallergy Research Laboratories of Savannah, Inc., Savannah, Georgia
  - Rush Presbyterian - St. Luke's Medical Center Rush University, Chicago, Illinois
  - South Bend Clniic, South Bend, Indiana
  - Clinical Research Specialist, Metairie, Louisiana
  - Doctor's Care, New Orleans, Louisiana
  - Children's International Medical Research, Slidell, Louisiana
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Heartland Clinical Research Inc., Omaha, Nebraska
  - Asthma & Allergy Center PC, Papillion, Nebraska
  - Office of Yekaterina Khronusova, MD, Las Vegas, Nevada
  - Pulmonary Medical Research of NY, PLLC, Bay Shore, New York
  - Asthma & Allergy Associates PC, Cortland, New York
  - AAIR Research Center, Rochester, New York
  - Office or Richard Castaldo, MD, Tonawanda, New York
  - Charlotte Lung and Health Center, Charlotte, North Carolina
  - Albermarle Allergy & Asthma PC, Elizabeth City, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - New Horizons Clinical Research, Inc., Cincinnati, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy Associates Research Center, LLC, Portland, Oregon
  - Valley Clinical Research Center, Easton, Pennsylvania
  - Advanced Clinical Concepts, Temple, Pennsylvania
  - Allergic Disease & Asthma Center PA, Greenville, South Carolina
  - Allergy & Asthma Consultants, LLP, Mt. Pleasant, South Carolina
  - Allergy and Asthma Clinic of Central Texas, Austin, Texas
  - Research Across America, Dallas, Texas
  - Breco Research, Houston, Texas
  - Breath of Life Research Institute, Houston, Texas
  - Lung Diagnostics, San Antonio, Texas
  - PI - Coor Clinical Research, LLC, Burke, Virginia
  - Pulmonary Associates of Richmond, inc., Richmond, Virginia
  - Rockwood Clinics, PS, Spokane, Washington
  - Allergy, Asthma and Sinus Center F.C., Greenfield, Wisconsin
  - Allergic Diseases, SC, West Allis, Wisconsin

REFERENCES:
- [Derived] Duan QL, Gaume BR, Hawkins GA, Himes BE, Bleecker ER, Klanderman B, Irvin CG, Peters SP, Meyers DA, Hanrahan JP, Lima JJ, Litonjua AA, Tantisira KG, Liggett SB. Regulatory haplotypes in ARG1 are associated with altered bronchodilator response. Am J Respir Crit Care Med. 2011 Feb 15;183(4):449-54. doi: 10.1164/rccm.201005-0758OC. Epub 2010 Sep 17. PMID 20851928
- See also: Patient's Instructions for Use — http://www.xopenex.com/about/patient-instructions.html